CLINICAL TRIAL: NCT00561340
Title: Caloric Supplementation During Long-Term Pharmacological Treatment of ADHD in Young Children
Brief Title: Study of the Effect of Calorie Supplementation on Growth in Young Children on ADHD Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0356-05-FB; B4Z-US-X018 (Other: Eli Lilly and Company); 11112 (Other: Abbott Laboratories)
Record Dates: First submitted 2007-11-16; First posted 2007-11-20 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: ADHD
Keywords: ADHD; Growth; Atomoxetine; Pediasure
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 Can of Pediasure Supplement Plus Nutritional Counseling (Experimental): Pediasure and nutritional counseling
  Interventions: Dietary Supplement: Pediasure; Behavioral: Nutritional counseling
- Counseling by the Provider on Ways to Encourage Caloric Intake (Active Comparator): Behavioral intervention - Nutritional Counseling
  Interventions: Behavioral: Nutritional counseling

INTERVENTIONS:
Dietary Supplement: Pediasure — 50% will be randomized to pediasure with nutritional counseling
  Arms: 1 Can of Pediasure Supplement Plus Nutritional Counseling
Behavioral: Nutritional counseling — 50% randomized to nutritional counseling only

SUMMARY:
The purpose of this study is to see if supplementing calories with Pediasure is effective in maintaining height, weight, and BMI percentiles for young children during 2 years of treatment with ADHD medication.

DETAILED DESCRIPTION:
This is a pilot study evaluating the effect of caloric supplementation on maintenance of growth parameters during two years of open-label atomoxetine treatment in 5 and 6 year old children with ADHD. The study will assess the efficacy of caloric supplementation in maintaining baseline percentiles for height, weight, and body mass index (BMI). Patients will be randomly assigned to receive either PediaSure for caloric supplementation, or no supplementation.

Secondary aims include assessing the tolerability and efficacy of long-term, open-label atomoxetine treatment in 5 and 6 year old children with ADHD, and obtaining adequate pilot data regarding the safety, efficacy, and potential effects of atomoxetine on growth parameters in order to submit a multisite R01 to more adequately assess atomoxetine treatment and its effects in young children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Children who participated in the 8 week DBPC trial of atomoxetine (1K23MH066127) who wish to participate in a long-term, open label trial of atomoxetine.
* Parents and patients must be able to attend regular study visits. Visits will be scheduled every 30 days for the first 6 months and then every 60 days for the next 18 months.
* Children who are on alternate medications due to inefficacy or intolerability of atomoxetine may still participate.

Exclusion Criteria:

* Parents who are unwilling to provide informed consent.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2006-01-02 (Actual); Primary Completion 2010-09-01 (Actual); Study Completion 2010-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Kratochvil, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Department of Psychiatry, Omaha, Nebraska, United States

REFERENCES:
- [Background] Spencer TJ, Newcorn JH, Kratochvil CJ, Ruff D, Michelson D, Biederman J. Effects of atomoxetine on growth after 2-year treatment among pediatric patients with attention-deficit/hyperactivity disorder. Pediatrics. 2005 Jul;116(1):e74-80. doi: 10.1542/peds.2004-0624. PMID 15995021

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 33 subjects total were eligible for participation in this study. 29 were enrolled and are included in the analysis. All patients had previously completed an 8-week double-blind placebo-controlled study of atomoxetine for the treatment of ADHD in 5 and 6 year olds.
Pre-assignment Details: 25 subjects were randomized to one of the 2 treatment groups. An additional 4 subjects for whom randomization to caloric supplementation was inappropriate were included in the nutritional counseling only arm for purposes of analysis as they did enroll in this study.
Period: Overall Study
Arm/Group | 1 Can of Pediasure Supplement Plus Nutritional Counseling | Counseling by the Provider on Ways to Encourage Caloric Intake
Started | 13 | 16
Completed | 7 | 16
Not Completed | 6 | 0
Not completed — refused to drink pediasure | 6 | 0

BASELINE CHARACTERISTICS:
Population: A total of 25 subjects were eligible for randomization. 4 subjects were not appropriate for randomization to caloric supplementation with pediasure so were included in the counseling only arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Can of Pediasure Supplement Plus Nutritional Counseling | Counseling by the Provider on Ways to Encourage Caloric Intake | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 16 | 29
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 8 | 11 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 12 | 15 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 11 | 12 | 23
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 16 | 29
ADHD treatment status [Number; unit: participants]
  Prior Active ADHD Treatment | 8 | 6 | 14
  Prior Placebo Treatment | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Description: Change in weight observed from baseline to 6 months
Time Frame: 6 months
Population: 29 of 33 eligible subjects were enrolled. 4 subjects were not eligible for randomization as they were not appropriate candidates for caloric supplementation. Of the 13 randomized to Pediasure, 6 subjects refused to drink it. Data is presented for any subject who drank any Pediasure.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | 1 Can of Pediasure Supplement Plus Nutritional Counseling | Counseling by the Provider on Ways to Encourage Caloric Intake
Number analyzed (Participants) | 13 | 16
kilograms | 0.37 (0.54) | -0.04 (0.33)

2. Primary Outcome: Height Change
Description: Change in height from baseline to 6 months
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | 1 Can of Pediasure Supplement Plus Nutritional Counseling | Counseling by the Provider on Ways to Encourage Caloric Intake
Number analyzed (Participants) | 13 | 16
centimeters | 1.85 (0.31) | 1.96 (0.44)

ADVERSE EVENTS:
Time Frame: Study duration was 2 years. Intervention (pediasure) was only during first 6 months of the study.
Description: Adverse events solicited through open-ended questioning of the parent and subject by the investigator
Arm/Group | 1 Can of Pediasure Supplement Plus Nutritional Counseling | Counseling by the Provider on Ways to Encourage Caloric Intake
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/16
Other Adverse Events (participants affected / at risk) | 0/13 | 0/16

LIMITATIONS AND CAVEATS:
This is a follow-up study of 5 and 6 year olds who completed a DBPC study of atomoxetine for ADHD. Data is confounded by subjects having entered the study on different pre-study and concurrent pharmacotherapy. The population is small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No